## TELEYOGA FOR CHRONIC LOW BACK PAIN: A QUANTITATIVE AND QUALITATIVE STUDY

## Sample size, statistical methods, and power calculation

Sample size: Based on the prior studies of tele-yoga (Table 1 and 2), sample size range is from 10 - 212 participants. The primary focus of this study being a feasibility trial, we propose to include n=20/group. Assuming 20% drop out rate, we plan to enroll 40 participants. We will report descriptive statistics for all who consent (including those who drop out) and for both groups with mean±SD for continuous variable and frequency (%) for categorical variables.

For Aim 1, Acceptability will use a paired t-test would be used to measure AIM<sup>1</sup> and semi structured qualitative interviews.

For Aim 2, paired t-test would be used to measure VAS, ODI, and PROMIS from prior to intervention and at 2 weeks as well as prior to intervention and 4 weeks.

For Aim 3, paired t-test would be used to measure FM2016, BAI, BDI from prior to intervention and at 2 weeks as well as prior to intervention and 4 weeks.